CLINICAL TRIAL: NCT01330043
Title: Extended Treatment for Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sean P. David, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU-09272010-6949; R01DA017441 (NIH); NCT01067612 (obsolete NCT alias)
Record Dates: First submitted 2010-10-07; First posted 2011-04-06 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Smoking Cessation
Keywords: smoking cessation intervention
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion; Tobacco Use Cessation Devices; Varenicline

STUDY DESIGN:
Intervention Model Description: Participants were randomized to extended or non-extended treatment and followed for 104 weeks.
Who Masked: Care Provider, Investigator
Masking Description: Behavioral therapists were blinded until the end of open-label treatment (26 weeks). Investigators were blinded to treatment assignment until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-extended treatment (Active Comparator): * 26 weeks of CBT
  * 10 weeks of combination bupropion plus nicotine patch
  * Additional 16 weeks of bupropion plus nicotine patch if increased craving or depression scores or varenicline if smoking at 10 weeks
  Interventions: Drug: Bupropion; Drug: Nicotine patch; Drug: Varenicline
- Extended treatment (Experimental): * 26 weeks of CBT
  * 10 weeks of combination bupropion plus nicotine patch
  * Additional 16 weeks of bupropion plus nicotine patch if increased craving or depression scores or varenicline if smoking at 10 weeks
  * 24 additional weeks of CBT
  Interventions: Drug: Bupropion; Drug: Nicotine patch; Drug: Varenicline

INTERVENTIONS:
Drug: Bupropion — Both groups received the same pharmacotherapy per protocol. During open label treatment, all received CBT and bupropion and NRT patch. At week 10 those who continued to smoke were switched to varenicline through week 26. At week 10 those who are abstinent and reported low levels of craving and low levels of depression symptoms were withdrawn from study medications. Those who were abstinent but reported difficulty with craving or depression symptoms remained on bupropion and NRT through week 26. Medication was not available after week 26.
  Other Names: Zyban
Drug: Nicotine patch — Both groups received the same pharmacotherapy per protocol. During open label treatment, all received CBT and bupropion and NRT patch. At week 10 those who continued to smoke were switched to varenicline through week 26. At week 10 those who are abstinent and reported low levels of craving and low levels of depression symptoms were withdrawn from study medications. Those who were abstinent but reported difficulty with craving or depression symptoms remained on bupropion and NRT through week 26. Medication was not available after week 26.
  Other Names: NRT
Drug: Varenicline — Both groups received the same pharmacotherapy per protocol. During open label treatment, all received CBT and bupropion and NRT patch. At week 10 those who continued to smoke were switched to varenicline through week 26. At week 10 those who are abstinent and reported low levels of craving and low levels of depression symptoms were withdrawn from study medications. Those who were abstinent but reported difficulty with craving or depression symptoms remained on bupropion and NRT through week 26. Medication was not available after week 26.
  Other Names: Chantix

SUMMARY:
Adult smokers (21-65) and adolescent smokers (18 - 21) years of age residing in Alameda and Santa Clara counties will serve as the target population for this study. A total of 400 smokers meeting eligibility criteria will be randomized. Treatment will include both open label and extended treatment phases. Randomization. Participants will be randomized to extended therapy or control conditions at baseline (prior to open label treatment) and the analysis will be intention-to-treat (ITT) to avoid the threat of selection bias. Primary hypothesis. Smokers randomized to receive CBT during extended treatment will have a higher prolonged abstinence rate (PA) at 52 week and 104 week follow-up than participants in the Supportive therapy Control treatment.

DETAILED DESCRIPTION:
During open label treatment, all receive CBT and bupropion and nicotine patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and nicotine replacement therapy (NRT) through week 26. Medication will not be available after week 26. All will receive CBT through week 26.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years at the beginning of the study Smoking at least 10 cigarettes a day (1/2 pack)

Exclusion Criteria:

1. Currently pregnant
2. Currently breastfeeding
3. Currently diagnosed with a seizure disorder, major depression, liver disease, kidney disease, congestive heart failure or diabetes mellitus
4. History of a seizure, seizure disorder, significant head trauma or central nervous system tumor
5. Family history of seizures
6. Currently using intravenous drugs
7. Currently using any drugs (marijuana, alcohol, cocaine, opiates, stimulants, etc.) on a daily basis
8. Currently using any over-the-counter stimulants and anorectics (diet pills)
9. Currently on bupropion (Wellbutrin, Wellbutrin SR) or other antidepressants, monoamine oxidase inhibitors, antipsychotics, benzodiazepines, theophylline, systemic steroids or levodopa
10. Currently on NRT or bupropion (Zyban)
11. Current or past diagnosis of anorexia nervosa or bulimia nervosa
12. Previous allergic response to bupropion or NRT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. David, MD, DPhil, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leyro TM, Crew EE, Bryson SW, Lembke A, Bailey SR, Prochaska JJ, Henriksen L, Fortmann SP, Killen JD, Killen DT, Hall SM, David SP. Retrospective analysis of changing characteristics of treatment-seeking smokers: implications for further reducing smoking prevalence. BMJ Open. 2016 Jun 29;6(6):e010960. doi: 10.1136/bmjopen-2015-010960. PMID 27357195
- [Result] Laude JR, Bailey SR, Crew E, Varady A, Lembke A, McFall D, Jeon A, Killen D, Killen JD, David SP. Extended treatment for cigarette smoking cessation: a randomized control trial. Addiction. 2017 Aug;112(8):1451-1459. doi: 10.1111/add.13806. Epub 2017 May 2. PMID 28239942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult cigarette smokers (N = 223) between the ages of 18 and 65 who smoked at least 10 cigarettes per day were included. Participants were randomized between 06/1/2010 and 01/22/2013.
Pre-assignment Details: Two participants were withdrawn from the study, of which one withdrew following a medication side effect of tachycardia and one participant was removed from the study for disruptive behavior -- both prior to randomization.
Groups:
- Maintenance Therapy: Participants will receive six months (26 weeks) of cognitive behavioral therapy (maintenance treatment) and a monthly phone call after 26 weeks asking about their smoking status and will not receive any treatment.
- Extended Treatment: Participants will receive twelve months (52 weeks) of cognitive behavioral therapy.
Period: Overall Study
Arm/Group | Maintenance Therapy | Extended Treatment
Started | 111 | 112
Completed | 111 | 108
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Maintenance Treatment: Participants receive 26 weeks of cognitive behavioral therapy (maintenance treatment) followed by a monthly phone call asking about their smoking status and will not receive any additional behavioral treatment after 26 weeks. Cognitive behavior therapy (CBT): During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26. All will receive CBT through week 26.
- Extended Treatment: Participants receive 52 weeks of cognitive behavioral therapy (maintenance plus extended treatment). Cognitive behavior therapy (CBT): During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26. All will receive CBT through week 52.
- Total: Total of all reporting groups
Arm/Group | Maintenance Treatment | Extended Treatment | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 43 (12) | 43 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 68 | 66 | 134
Region of Enrollment [Number; unit: participants]
  United States | 111 | 112 | 223

OUTCOME MEASURES:

1. Primary Outcome: Expired-air CO Verified Point-prevalence Abstinence
Description: Self-reported no smoking in last 7 days verified by CO<10 ppm
Time Frame: 52 weeks
Measure: Number; unit: participants
Groups:
- Maintenance Treatment: Participants receive 26 weeks of cognitive behavioral therapy (maintenance treatment) followed by a monthly phone call asking about their smoking status and will not receive any additional behavioral treatment after 26 weeks. During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26. All will receive CBT through week 52.
- Extended Treatment: Participants receive 52 weeks of cognitive behavioral therapy (extended treatment). During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26. All will receive CBT through week 52.
Arm/Group | Maintenance Treatment | Extended Treatment
Number analyzed (Participants) | 111 | 108
participants | 44 | 42

2. Secondary Outcome: Expired-air CO Verified Point-prevalence Abstinence
Description: Self-reported no smoking in last 7 days verified by CO<10 ppm
Time Frame: 104 weeks
Measure: Number; unit: participants
Arm/Group | Maintenance Treatment | Extended Treatment
Number analyzed (Participants) | 111 | 108
participants | 39 | 33

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over 104 weeks.
Description: Participants were queried at every in-person visit for adverse events and asked to call the health educator if they developed any troubling side effects or medical events. All side effects or adverse events were reported to the study physician who provided clinical advice as needed.
Groups:
- Maintenance Treatment: Participants receive 26 weeks of cognitive behavioral therapy (maintenance treatment) followed by a monthly phone call asking about their smoking status and will not receive any additional behavioral treatment after 26 weeks. Cognitive behavior therapy (CBT): During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26.
  Maintenance treatment (cognitive behavioral therapy)(CBT): During open label treatment, all receive CBT and bupropion and NRT patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 1
- Extended Treatment: Participants receive 26 weeks of cognitive behavioral therapy (maintenance treatment) followed by another 26 weeks of cognitive behavioral therapy (extended treatment). Cognitive behavior therapy (CBT): During open label treatment, all receive CBT and bupropion and nicotine replacement therapy (NRT) patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of craving and low levels of depression symptoms will be withdrawn from study medications. Those who are abstinent but report difficulty with craving or depression symptoms will remain on zyban and NRT through week 26.
  Maintenance treatment (cognitive behavioral therapy)(CBT): During open label treatment, all receive CBT and bupropion and NRT patch. At week 10 those who continue to smoke will be switched to varenicline through week 26. At week 10 those who are abstinent and report low levels of cravin
Arm/Group | Maintenance Treatment | Extended Treatment
All-Cause Mortality (participants affected / at risk) | 0/111 | 2/112
Serious Adverse Events (participants affected / at risk) | 0/111 | 3/112
Other Adverse Events (participants affected / at risk) | 22/111 | 20/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Treatment (N=111) | Extended Treatment (N=112)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Rapid heart rate associated with syncopal or near-syncopal event
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Death from lung cancer during the follow-up period
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Death from myocardial infection during the follow-up period
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Treatment (N=111) | Extended Treatment (N=112)
Anxiety (Psychiatric disorders) | 11 (11) | 8 (8)
Dry mouth (General disorders) | 15 (15) | 11 (11)
Headache (Nervous system disorders) | 6 (6) | 9 (9)
Insomnia (Nervous system disorders) | 16 (16) | 13 (13)
Nausea (Gastrointestinal disorders) | 9 (9) | 4 (4)
Vivid dreams (Nervous system disorders) | 22 (22) | 20 (20)

LIMITATIONS AND CAVEATS:
The target sample size of N=400 was not reached due to challenges with recruitment, however, the sample size achieved was sufficient to test main effects of extended treatment on abstinence outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No